CLINICAL TRIAL: NCT05600959
Title: The Role of Cytokines in Early Diagnosis, Assessment of Response and Prognosis of Patients With Lymphoma-associated Hemophagocytic Lymphohistiocytosis
Brief Title: Sensitivity and Specificity of Cytokines in the Diagnosis of Lymphoma-associated HLH
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Beijing Friendship Hospital (Other)
Responsible Party: Principal Investigator, Zhao Wang, Professor and Head of hematology, Beijing Friendship Hospital
Other Study IDs: BFH20221009001/BFHHZML20220006
Record Dates: First submitted 2022-10-27; First posted 2022-11-01 (Actual); Last update posted 2022-11-01 (Actual); Status verified 2022-10

CONDITIONS: Hemophagocytic Lymphohistiocytoses; Lymphoma
Keywords: Hemophagocytic Lymphohistiocytosis; Lymphoma; Cytokine; Diagnosis
MeSH Terms: conditions — Lymphohistiocytosis, Hemophagocytic; Lymphoma; Disease | interventions — Th1-Th2 Balance

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Lymphoma group: Patients with histopathologically confirmed lymphoma who did not receive systemic chemotherapy before enrollment.
  Interventions: Diagnostic Test: cytokine
- Lymphoma-associated HLH group: Patients with histopathologically confirmed lymphoma who meet HLH-04 diagnostic criteria, and did not receive systemic chemotherapy before enrollment.
  Interventions: Diagnostic Test: cytokine

INTERVENTIONS:
Diagnostic Test: cytokine — Peripheral blood samples were collected at diagnosis, 2 weeks after the first cycle of chemotherapy and 2 weeks after the second cycle of chemotherapy to monitor cytokine level changes.

SUMMARY:
Lymphoma-associated hemophagocytic lympohistiocytosis is a refractory immune disorder with high mortality. Early identification and diagnosis of lymphoma-associated HLH has become the key to improve the prognosis of lymphoma-associated HLH. Therefore, we conduct a multicenter, prospective, observational clinical study to explore the sensitivity and specificity of cytokines for the early diagnosis of lymphoma-associated HLH.

DETAILED DESCRIPTION:
Lymphoma-associated hemophagocytic lympohistiocytosis is a refractory immune disorder with high mortality. Without early intervention, the median survival time is less than 2 months. Early identification and diagnosis of lymphoma-associated HLH has become the key to improve the prognosis of lymphoma-associated HLH. Therefore, it is urgent to find a method for the early diagnosis of lymphoma-associated HLH. We conduct a multicenter, prospective, observational clinical study to explore the sensitivity and specificity of cytokines for the early diagnosis of lymphoma-associated HLH, and its correlation with disease severity, treatment response, and prognosis.

ELIGIBILITY:
Inclusion Criteria:

* Age 40-75, gender is not limited.
* Patients with histopathologically confirmed lymphoma who meet HLH-04 diagnostic criteria, and did not receive systemic chemotherapy before enrollment.
* Patients with histopathologically confirmed lymphoma who did not receive systemic chemotherapy before enrollment.
* Informed consent obtained.

Exclusion Criteria:

* Patients with severe active infections (viral, bacterial, fungal, or parasitic).
* Patients with active autoimmune disease or a history of organ transplantation who are receiving immunosuppressive therapy.
* Patients with other type of malignant tumors within 5 years, except for cured solid tumors.
* Patients planned to receive immunotherapy.
* Pregnant and breastfeeding females.
* History of human immunodeficiency virus (HIV) infection.
* Acute or chronic active hepatitis B or hepatitis C.
* Patients assessed as ineligible for the study by the investigator.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with lymhoma and patients with lymphoma-associated HLH
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2022-11-01 (Estimated); Primary Completion 2025-11-01 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
The sensitivity and specificity of cytokines to predict lymphoma-associated HLH | 1 year
  The sensitivity and specificity of cytokines as a means of early diagnosis of lymphoma-associated hemophagocytic lymphohistiocytosis

SECONDARY OUTCOMES:
Dynamic changes of cytokine levels during treatment | 1 years
  To monitor the correlation between cytokine levels and disease severity, treatment response and prognosis of lymphoma-associated hemophagocytic lymphohistiocytosis

CONTACTS AND LOCATIONS:
Overall Officials: Zhao Wang, MD, Principal Investigator — Beijing Friendship Hospital
Locations (1):
- Zhao Wang, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No